CLINICAL TRIAL: NCT01864174
Title: A 24-Week International, Multi-center, Randomized, Parallel-group, Double-blind Trial to Evaluate Metformin Extended Release Monotherapy Compared to Metformin Immediate Release Monotherapy in Adults Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise
Brief Title: Phase 4: Investigational Study to Evaluate Metformin XR Monotherapy Versus Metformin IR Monotherapy in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-206; 2012-004531-23 (EudraCT Number)
Record Dates: First submitted 2013-05-24; First posted 2013-05-29 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Metformin XR and Placebo matching with Metformin XR (Active Comparator): Metformin Extended Release (XR) 500 mg tablets (500-2000 mg per day) by mouth twice daily (BID) for 24 weeks
  Placebo matching with Metformin XR 0 mg tablets by mouth twice daily (BID) for 24 weeks
  Interventions: Drug: Metformin XR; Drug: Placebo matching with Metformin XR
- Arm 2: Metformin IR and Placebo matching with Metformin IR (Active Comparator): Metformin Immediate Release (IR) 500 mg tablets (500-2000 mg per day) by mouth twice daily (BID) for 24 weeks
  Placebo matching with Metformin IR 0 mg tablets by mouth twice daily (BID) for 24 weeks
  Interventions: Drug: Metformin IR; Drug: Placebo matching with Metformin IR

INTERVENTIONS:
Drug: Metformin XR
  Other Names: Glucophage XR
  Arms: Arm 1: Metformin XR and Placebo matching with Metformin XR
Drug: Metformin IR
  Other Names: Glucophage
  Arms: Arm 2: Metformin IR and Placebo matching with Metformin IR
Drug: Placebo matching with Metformin XR
  Arms: Arm 1: Metformin XR and Placebo matching with Metformin XR
Drug: Placebo matching with Metformin IR
  Arms: Arm 2: Metformin IR and Placebo matching with Metformin IR

SUMMARY:
The purpose of this study is determine if Metformin XR monotherapy in subjects with type 2 diabetes is non-inferior to Metformin IR monotherapy

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women, aged ≥18 years old at time of enrollment
* Treatment naive subjects with type 2 diabetes mellitus with inadequate glycemic (HbA1c ≥7.0% and ≤9.2% obtained at screening visit) control on diet and exercise alone
* Women must have a negative serum or urine test within 24 hours prior to start of investigational product

Exclusion Criteria:

* History of ketoacidosis, lactic acidosis or hyperosmolar non-ketonic coma
* Symptoms of poorly controlled diabetes, including but not limited to marked polyuria and polydipsia with >10% weight loss during last 3 months
* Serum creatinine ≥1.50 mg/dL (133 μmol/L) for male subjects; serum creatinine ≥1.40 mg/dL (124 μmol/L for female subjects)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1736 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (133):
- United States (38):
  - Central Alabama Research, Birmingham, Alabama
  - Terence T. Hart, Md, Muscle Shoals, Alabama
  - Clini Res Advantage Desert Clin Res, Llc, Mesa, Arizona
  - Clinical Res Advantage Central, Phoenix, Arkansas
  - Marin Endocrine Care And Research, Inc., Greenbrae, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Actca, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - R. Srinivasan, M.D., Inc., Monterey Park, California
  - Diabetes Medical Center Of California, Northridge, California
  - Valley Clinical Trials, Northridge, California
  - Center For Clinical Trials Of Sacramento, Inc., Sacramento, California
  - Clinical Research Advantage, Colorado Springs, Colorado
  - Colorado Springs Family Practice, Colorado Springs, Colorado
  - Clinical Research Advantage, Inc/Co Springs Health Partners, Briar, Colorado Springs, Colorado
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Family Care Partners, Jacksonville, Florida
  - Omega Research Consultants, Llc, Orlando, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Gulfcoast Medical Research Center, Llc, Tampa, Florida
  - Cedar-Crosse Research Ctr, Chicago, Illinois
  - Clinical Research Advantage, Inc./Family Medicine Associates, Evansville, Indiana
  - American Health Network Of In Llc, Muncie, Indiana
  - Columbia Medical Practice, Columbia, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Drs. Rodbard And Dempsey, Rockville, Maryland
  - Ny Clinical Trials, New York, New York
  - White Oak Family Physicians, Pa, Asheboro, North Carolina
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Medical Research Unlimited, Inc., Cincinnati, Ohio
  - Lion Research, Norman, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Integrated Medical Group Pc / Fleetwood Medical Assoc., Fleetwood, Pennsylvania
  - Palmetto Clinical Trial Services Llc, Fountain Inn, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Covenant Clinical Research, Pa, San Antonio, Texas
  - Independence Family Medicine, Virginia Beach, Virginia
- Canada (10):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Brampton, Ontario
  - Local Institution, Burlington, Ontario
  - Local Institution, Collingwood, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Newmarket, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Québec, Quebec
  - Local Institution, London
- Czechia (8):
  - Local Institution, Brno
  - Local Institution, České Budějovice
  - Local Institution, Krnov
  - Local Institution, Liberec
  - Local Institution, Litomyšl
  - Local Institution, Nový Jičín
  - Local Institution, Ostrava-Kunčice
  - Local Institution, Prague
- Germany (10):
  - Local Institution, Aschaffenburg, Bavaria
  - Local Institution, Münster, North Rhine-Westphalia
  - Local Institution, Leipzig, Saxony
  - Local Institution, Berlin
  - Local Institution, Heidelberg
  - Local Institution, Leipzig
  - Local Institution, Löhne
  - Local Institution, Myen
  - Local Institution, Papenburg
  - Local Institution, Pirna
- Hungary (15):
  - Local Institution, Pécs, Baranya
  - Local Institution, Szigetvár, Baranya
  - Local Institution, Sátoraljaújhely, Borsod-Abauj Zemplen county
  - Local Institution, Hodmezvasarhely, Csongrád megye
  - Local Institution, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Local Institution, Budapest
  - Local Institution, Csorna
  - Local Institution, Debrecen
  - Local Institution, Kecskemét
  - Local Institution, Mosonmagyaróvár
  - Local Institution, Nagykanizsa
  - Local Institution, Orosháza
  - Local Institution, Szentes
  - Local Institution, Székesfehérvár
  - Local Institution, Szobathely
- Poland (7):
  - Local Institution, Gdansk, Pomeranian Voivodeship
  - Local Institution, Katowice, Silesian Voivodeship
  - Local Institution, Bialystok
  - Local Institution, Krakow
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Zamość
- Puerto Rico (14):
  - Local Institution, Caguas, PR
  - Local Institution, Carolina, PR
  - Local Institution, Río Grande, PR
  - Local Institution, Las Lomas, San Juan
  - Luis Rivera-Colon, Md, Las Lomas, San Juan
  - Fb Med Research, Psc, Caguas
  - Policlinica Dr. Luis Rodriguez, Carolina
  - Local Institution, Ponce
  - Ponce School Of Medicine, Ponce
  - Research & Cardiovascular Corp, Ponce
  - Caparra Internal Med Res Ctr, Río Grande
  - Altamira Family Medicine And Research Institute, San Juan
  - Local Institution, San Juan
  - The Office Of Miguel Sosa-Padilla, Md, San Juan
- Romania (9):
  - Local Institution, Alba Iulia
  - Local Institution, Bacau
  - Local Institution, Baia Mare
  - Local Institution, Brasov
  - Local Institution, Bucharest
  - Local Institution, Constanța
  - Local Institution, Ploieşti
  - Local Institution, Satu Mare
  - Local Institution, Tg Mures
- South Africa (11):
  - Local Institution, Mthatha, Eastern Cape
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Welkom, Free State
  - Local Institution, Lyttelton, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Phoenix, Durban, KwaZulu-Natal
  - Local Institution, Brits, North West
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Worcester, Western Cape
  - Local Institution, Potchefstroom
- United Kingdom (11):
  - Local Institution, Monifieth, AFO
  - Local Institution, Carmarthen, CAT
  - Local Institution, Fife, FIF
  - Local Institution, Chippenham, Wiltshire
  - Local Institution, Chippenham, WLT
  - Local Institution, Addlestone
  - Local Institution, Bath
  - Local Institution, Cardenden Fife
  - Local Institution, Dundee
  - Local Institution, Manchester
  - Local Institution, Nuneaton

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS clinical trial educational resource — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1736 enrolled at 148 study sites in North America, Europe, and South Africa.Lead in period=794. Reasons not entered: 1 AE, 17 WC, 4 lost to FU, 3 NC, 911 SC, 4 ARS, 1 other. Adverse event=-AE, Withdrew consent=WC, Follow-up=FU, poor/non-compliance=NC, No longer met study criteria=SC, Administrative reason by sponsor=ARS.
Pre-assignment Details: 570 completed lead-in period and were eligible for randomization. 568 randomized. Non-randomized: 1 AE, 27 WC, 3 lost to FU, 7 NC, 159 SC, 8 ARS, 3 other.
Groups:
- Metformin XR: Participants received Metformin XR and Placebo matching with Metformin XR
  Metformin Extended Release (XR) 500 mg tablets (500-2000 mg per day) by mouth twice daily (BID) for 24 weeks
  Placebo matching with Metformin XR 0 mg tablets by mouth twice daily (BID) for 24 weeks.
- Metformin IR: Participants received Metformin IR and Placebo matching with Metformin IR.
  Metformin Immediate Release (IR) 500 mg tablets (500-2000 mg per day) by mouth twice daily (BID) for 24 weeks
  Placebo matching with Metformin IR 0 mg tablets by mouth twice daily (BID) for 24 weeks.
Period: Double Blind Treatment - All Treated
Arm/Group | Metformin XR | Metformin IR
Started | 283 | 285
Completed | 268 | 271
Not Completed | 15 | 14
Not completed — Removed due to site non-compliance | 15 | 14
Period: Double Blind - Compliant Randomized
Arm/Group | Metformin XR | Metformin IR
Started | 268 | 271
Completed | 245 | 245
Not Completed | 23 | 26
Not completed — Adverse Event | 6 | 1
Not completed — Subject Request to Discontinue Treatment | 2 | 0
Not completed — Subject Withdrew Consent | 4 | 5
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 10
Not completed — Poor/Non-compliance | 1 | 0
Not completed — Other | 6 | 10
Period: Off Treatment Follow-Up
Arm/Group | Metformin XR | Metformin IR
Started | 9 | 1
Completed | 6 | 1
Not Completed | 3 | 0
Not completed — Other | 2 | 0
Not completed — Subject Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Data Set (n=568) are the randomized participants who received at least 1 dose of study drug during the double blind treatment period (up to rescue). 29 participants were excluded from the baseline Randomized Data Set; therefore, the number of participants included in the baseline population is 539. n = number of evaluable participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin XR | Metformin IR | Total
Number analyzed (Participants) | 268 | 271 | 539
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.69) | 55.3 (10.34) | 56.0 (10.53)
Age, Customized [Number; unit: participants]
  < 65 years | 198 | 226 | 424
  >= 65 years | 70 | 45 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 122 | 244
  Male | 146 | 149 | 295
Race/Ethnicity, Customized [Number; unit: participants]
  White | 227 | 225 | 452
  Black or African American | 22 | 19 | 41
  Asian | 17 | 20 | 37
  Other | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in HbA1c
Description: Mean change in glycated hemoglobin (HbA1c) from baseline to Week 24 in the double-blind treatment period.
Time Frame: Baseline and Week 24
Population: Randomized participants who took at least one dose of double-blind study medication in the treatment group to which they were randomized with non-missing baseline and Week 24 values who were not excluded due to non-compliance.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Metformin XR | Metformin IR
Number analyzed (Participants) | 237 | 237
percent | -0.93 (0.0485) [-1.02 to -0.83] | -0.96 (0.0480) [-1.05 to -0.87]
Statistical Analysis 1: Comparison: Metformin XR vs Metformin IR; Test type: Non-Inferiority or Equivalence — The study provided 90% power to demonstrate noninferiority in change from baseline mean HbA1c at Week 24, with an assumed standard deviation (SD) of 1.0%, a non-inferiority margin of 0.3%, and 2-sided alpha of 0.05 for the primary comparison; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.10 to 0.17], Standard Error of Mean 0.0687 — METFORMIN XR VS METFORMIN IR

2. Secondary Outcome: Mean Change in Fasting Plasma Glucose (FPG)
Description: The mean change in fasting plasma glucose (FPG) from baseline to Week 24 in the double-blind treatment period was assessed. The lack of glycemic control criteria for initiation of rescue medication during Week 12 to Week 24 was having a FPG > 200 mg/dL (11.1 mmol/L). mg/dL = milligrams per deciliter; mmol/L = millimole per Liter
Time Frame: Baseline and Week 24
Population: Randomized participants who took at least one dose of double-blind study medication in the treatment group to which they were randomized with non-missing baseline and Week 24 values and who were not excluded due to non-compliance.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Metformin XR | Metformin IR
Number analyzed (Participants) | 228 | 229
mg/dL | -21.1 (1.803) | -20.6 (1.789)

3. Secondary Outcome: Mean Change in Mean Daily Glucose (MDG)
Description: The mean change in Mean Daily Glucose (MDG) from baseline to Week 24 in the double-blind treatment period was assessed. Prior to the Day 1 visit (between Week -1 and Day 1) and in the week before the Week 24/Study Termination and Rescue or Early Treatment Termination visit, participants performed 7-point finger stick blood glucose monitoring (before and 2 hours after 3 meals per day, and at bedtime) for 3 consecutive days in order to determine their MDG.
Time Frame: Baseline and Week 24
Population: Randomized participants who took at least one dose of double-blind study medication in the treatment group to which they were randomized with non-missing baseline and Week 24 last observation carried forward (LOCF) results who were not excluded due to non-compliance.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Metformin XR | Metformin IR
Number analyzed (Participants) | 211 | 218
mg/dL | -24.68 (1.5813) | -27.05 (1.555)

4. Secondary Outcome: Percent of Participants With HbA1c < 7%
Description: Percent of participants achieving a therapeutic glycemic response (defined as HbA1c < 7.0%) at Week 24 in the double-blind treatment period.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Metformin XR | Metformin IR
Number analyzed (Participants) | 237 | 237
percent of participants | 70.9 [65.5 to 76.3] | 72.0 [66.3 to 77.7]

5. Primary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), SAEs Related to Study Therapy, SAEs Leading to Discontinuation, Adverse Events (AEs) Related to Study Therapy, and AEs Leading to Discontinuation
Description: SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Treatment-related=having certain, probable, possible, or missing relationship to study drug. All listed events are treatment emergent, which is defined as nonserious and serious AEs with an onset from Day 1 of the double-blind treatment up to and including 4 days and 30 days respectively, after the last dose date of double-blind study. randomized.
Time Frame: Date of first dose (Day 1) up to 30 post last dose of study drug (approx. 28 weeks)
Population: Treated participants; All participants who took at least one dose of double-blind study medication in the treatment group they were randomized to unless participants had never received the double-blind study medication they were randomized. Those participants were included in the treatment group based on the first treatment received.
Measure: Number; unit: participants
Arm/Group | Metformin XR | Metformin IR
Number analyzed (Participants) | 283 | 285
participants
  Death | 1 | 0
  SAE | 8 | 10
  SAEs Related to Study Therapy | 1 | 1
  SAEs Leading to Discontinuation | 0 | 1
  AEs Related to Study Therapy | 30 | 25
  AEs Leading to Discontinuation | 10 | 7

ADVERSE EVENTS:
Time Frame: From Day 1 up to 30 days post last dose (approx. 28 weeks)
Arm/Group | Metformin XR | Metformin IR
Serious Adverse Events (participants affected / at risk) | 8/283 | 10/285
Other Adverse Events (participants affected / at risk) | 25/283 | 22/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin XR (N=283) | Metformin IR (N=285)
Hypocoagulable state (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin XR (N=283) | Metformin IR (N=285)
Diarrhoea (Gastrointestinal disorders) | 25 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.